CLINICAL TRIAL: NCT00332553
Title: Study of Vasomotor Symptoms in Postmenopausal Women Receiving Combination Raloxifene and Oral Estrogen
Brief Title: Study of Hot Flashes and Night Sweats in Postmenopausal Women Receiving Combination Raloxifene and Oral Estrogen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 5546; H3S-US-GGKM
Record Dates: First submitted 2006-05-30; First posted 2006-06-01 (Estimated); Last update posted 2007-05-15 (Estimated); Status verified 2007-05

CONDITIONS: Vasomotor Symptoms; Endometrial Safety
MeSH Terms: interventions — Raloxifene Hydrochloride; Medroxyprogesterone Acetate; Estrogens; Estradiol

INTERVENTIONS:
Drug: Raloxifene
Drug: medroxyprogesterone acetate
Drug: estrogen
Drug: 17 beta estradiol

SUMMARY:
This pilot study was designed to explore the effects of combined treatment with raloxifene HCl 60 mg and oral 17 beta-estradiol 1mg/day on the number of vasomotor episodes (hot flashes plus night sweats) in postmenopausal women discontinuing continuous combined hormone replacement therapy (ccHRT) compared to women treated with raloxifene HCl 60 mg alone.

ELIGIBILITY:
Inclusion Criteria:

* Post menopausal women, 50-70 years of age
* Had taken ccHRT for at least 6 months prior to study entry
* No unexplained vaginal bleeding in the 3 months prior to study entry
* Understand and sign an informed consent document

Exclusion Criteria:

* Prior hysterectomy
* Endometrial thickness (excluding endometrial fluid) greater than 8 mm or endometrial fluid greater than or equal to 4 mm at study entry
* Abnormal Pap smear at study screening or within the preceding 3 years
* Abnormal transvaginal ultrasound result at study screening
* Past or current history of malignant neoplasms

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2002-02; Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
Compare the number of vasomotor symptoms at 12 weeks between those women taking the combination of raloxifene with oral estradiol versus those taking raloxifene alone.

SECONDARY OUTCOMES:
Determine the effect of treatment with combined raloxifene and estradiol compared with raloxifene alone on the severity of vasomotor symptoms as well as on the frequency and severity of hot flashes and night sweats
Determine the effects of treatment with combined raloxifene and estradiol in postmenopausal women on endometrial and general safety

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM-5PM Eastern time (UTC/GMT-5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877- CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Indianapolis, Indiana, United States